CLINICAL TRIAL: NCT07252687
Title: The Effect of Gender-affirmative Measures on Breast Perception in Trans Men (TRANSBREAST) - a Prospective Cohort Study
Brief Title: The Effect of Gender-affirmative Measures on Breast Perception in Trans Men
Acronym: TRANSBREAST
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1125/2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Transgender; Gender Dysphoria in Adolescents and Adults
Keywords: transgender; breastdysphoria; trans male; non binary; genderdiverse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: quality of life questionnaire- iTransQoL, chest dysphoria measure — Before starting treatment, participants should complete the Chest Dysphoria Measure and iTransQoL questionnaires (=time point 0). The second time point for completing the questionnaires again is 3 months after starting hormone therapy. Subsequently, the questionnaires should be completed a third time after breast-affirming surgery. The final survey takes place two years after time point 0, or 6 months after the previous survey.

SUMMARY:
Breast dysphoria in transmasculine or genderdiverse individuals is a distinct psychological burden associated with depression, anxiety and suicidality. The aim is to systematically investigate the effect of GAHT (gender-affirming hormone therapy) and mastectomy on this form of dysphoria.

The primary objective of this study is to analyse and investigate the psychological and physical effects of breast development on trans men or genderdiverse individuals.

A secondary objective is to determine the extent to which the stress affects the well-being of trans men depending on the coping strategies used (binding vs. taping).

ELIGIBILITY:
Inclusion Criteria:

* AFAB (Assigned Female At Birth)
* before starting GAHT
* before mastectomy

Exclusion Criteria:

* Ongoing GAHT
* Mastectomy already performed
* Lack of capacity to give consent
* Insufficient knowledge of German

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — trans men and gender diverse persons
Study Population: Referral to the medical University of Innsbruck Hospital or a cooperating center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Chest Dysphoria Measure Score | From enrollment to the end of observation after 2 years
  Chest Dysphoria Measure Score before GAHT, during GAHT, and after mastectomy